CLINICAL TRIAL: NCT03786354
Title: Prospective Evaluation of Shoulder Morbidity in Patients With Lymph-Node Positive Breast Cancer Receiving Regional Nodal Irradiation
Brief Title: Intensity Modulated Radiation Therapy or 3-Dimensional Conformal Radiation Therapy in Treating Patients With Lymph-Node Positive Breast Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Sasha Beyer, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSU-18201; NCI-2018-02307 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2018-12-19; First posted 2018-12-26 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Lymph Node Involvement; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8
MeSH Terms: interventions — Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arm A (IMRT) (Experimental): Patients undergo Intensity-Modulated Radiation Therapy over 5 weeks.
  Interventions: Radiation: Intensity-Modulated Radiation Therapy
- Arm B (3DCRT) (Experimental): Patients undergo 3-Dimensional Conformal Radiation Therapy over 5 weeks.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy

INTERVENTIONS:
Radiation: 3-Dimensional Conformal Radiation Therapy — Undergo 3DCRT
  Other Names: 3-dimensional radiation therapy; 3D CONFORMAL RADIATION THERAPY; 3D CRT; 3D-CRT; Conformal Therapy; Radiation Conformal Therapy
  Arms: Arm B (3DCRT)
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy
  Arms: Arm A (IMRT)

SUMMARY:
This phase II trial studies the shoulder morbidity in patients with lymph-node positive breast cancer receiving intensity modulated radiation therapy or 3-dimensional conformal radiation therapy. Intensity modulated radiation therapy may cause less shoulder/arm morbidity in patients with lymph-node positive breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if intensity modulated radiation therapy (IMRT) reduces average 1-year patient-reported shoulder/arm morbidity in women receiving regional nodal irradiation (RNI) for lymph-node positive breast cancer as compared to historical data.

SECONDARY OBJECTIVES:

I. To measure patient-reported shoulder/arm morbidity in women receiving RNI with 3-dimensional conformal radiation therapy (3DCRT) for lymph-node positive breast cancer.

II. To measure change in shoulder range of motion in women receiving RNI. III. To measures rates of ipsilateral upper extremity lymphedema in women receiving RNI.

IV. To explore the dose volume parameters to the shoulder/neck/trunk musculature associated with worsening patient-reported shoulder/arm morbidity.

V. To assess disease outcomes in patients treated with IMRT. VI. To measure long-term patient-reported shoulder/arm morbidity in women receiving RNI with IMRT or 3DCRT.

OUTLINE: Patients are assigned to 1 of 2 arms.

ARM A: Patients undergo IMRT over 5 weeks.

ARM B: Patients undergo 3DCRT over 5 weeks.

After completion study treatment, patients are followed up at 1, 6, and 12 months, and then annually for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven diagnosis of breast cancer
* Patients that receive neoadjuvant systemic therapy (chemotherapy, anti-HER2 therapy, or endocrine therapy) are eligible
* History/physical examination within 60 days prior to study entry
* Patients who have undergone either a lumpectomy or mastectomy are eligible
* Patients that have undergone any type of breast reconstruction are eligible
* The interval between the date of last surgery or chemotherapy and registration must be =< 84 days
* Women of childbearing potential must have a negative urine or serum pregnancy test within 14 days of start of radiation therapy
* Women of childbearing potential must be non-pregnant and non-lactating and willing to use medically acceptable form of contraception during radiation therapy
* Patients must provide study specific informed consent prior to study entry

Exclusion Criteria:

* Clinical or radiologic evidence of distant metastases
* Patients with known unresected disease in the axillary apex or supraclavicular fossa
* Prior invasive or in-situ carcinoma of the breast (prior lobular breast carcinoma in situ [LCIS] is eligible)
* Prior surgery to the ipsilateral shoulder for any condition
* Baseline impaired mobility of the ipsilateral shoulder from a condition not related to the breast cancer surgery as determined by the treating physician
* Non-epithelial breast malignancies such as sarcoma/lymphoma
* Prior radiotherapy to the breast or prior radiation to the region of the ipsilateral breast that would result in overlap of radiation fields
* Medical, psychiatric, or other conditions that would prevent the patient from receiving the protocol therapy or providing informed consent
* Pregnancy or women of childbearing potential who are sexually active and not willing/able to use medically acceptable forms of contraception
* Active systemic lupus, erythematosus, or any history of scleroderma, dermatomyositis with active rash

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Shoulder/arm morbidity assessed by Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire in patients treated with intensity modulated radiation therapy (IMRT) | At 1 year
  DASH questionnaire in patients treated with IMRT to assess shoulder/arm morbidity. Patients that have a DASH score of ≥15 at 1 year post-treatment will be considered as having persistent shoulder morbidity. The full scale range is 0-100.

SECONDARY OUTCOMES:
Shoulder/arm morbidity assessed by DASH questionnaire in patients treated with 3-dimensional conformal radiation therapy (3DCRT) | At 1 year
  DASH questionnaire in patients treated with 3DCRT to assess shoulder/arm morbidity. Patients that have a DASH score of ≥15 at 1 year post-treatment will be considered as having persistent shoulder morbidity.
Changes in shoulder range of motion for flexion, abduction, internal and external rotation using a goniometer as defined by the American Academy of Orthopedic Surgeons | At baseline, 1 month, 6 months and 12 months post-radiation
  Using a goniometer as defined by the American Academy of Orthopedic Surgeons to measure changes in shoulder range of motion for flexion, abduction, internal and external rotation
Measure rates of upper extremity lymphedema using arm circumference with a tape measure | At baseline, 1 month, 6 months and 12 months post-radiation
  Measure rates of upper extremity lymphedema using arm circumference using a tape measure
Measure rates of upper extremity lymphedema using a perometer | At baseline, 1 month, 6 months and 12 months post-radiation
  Measure rates of upper extremity lymphedema using arm circumference using a perometer
Dosimetric parameters associated with worse arm/shoulder morbidity as measured by the DASH | Up to 5 years
  Dosimetric parameters (the volume of shoulder receiving 5-50 Gy) associated with worse arm/shoulder morbidity as measured by the DASH
Rates of loco-regional control in patients treated with IMRT | At 5 years
  Rates of loco-regional control, distant metastases, and overall survival in patients treated with IMRT
Distant metastases in patients treated with IMRT | At 5 years
  The cumulative incidence of distant metastases at 5 years in patients treated with IMRT control, distant metastases
Overall survival in patients treated with IMRT | Up to 5 years
  Kaplan-Meier method will be used to estimate the 5-year overall survival in patients treated with IMRT
Shoulder/arm morbidity using the DASH questionnaire in patients treated with IMRT | Up to 5 years
  DASH questionnaire in patients treated with IMRT to assess shoulder/arm morbidity using full scale range 0-100
Shoulder/arm morbidity using the DASH questionnaire in patients treated with 3DCRT | Up to 5 years
  DASH questionnaire in patients treated with 3DCRT to assess shoulder/arm morbidity

CONTACTS AND LOCATIONS:
Overall Officials: Sasha Beyer, MD, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu